CLINICAL TRIAL: NCT00621166
Title: The Pharmacokinetics and Safety of Generic Lopinavir/Ritonavir (200/50 mg Tablets) 400/100 mg q12h in Thai HIV-infected Pregnant Women
Brief Title: Pharmacokinetics of Generic Lopinavir/Ritonavir in Pregnant Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIV-NAT 093; approved
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: Generic lopinavir/ritonavir; Pharmacokinetics; Pregnancy; Antiviral activity; Safety
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): generic lopinavir/ritonavir
  Interventions: Drug: generic lopinavir/ritonavir

INTERVENTIONS:
Drug: generic lopinavir/ritonavir — Patients will start with lopinavir/ritonavir new formulation 400/100 mg bid with a low fat diet plus 2 nucleoside reverse transcriptase inhibitors (NRTIs). The choice of the 2 NRTIs is at the discretion of the investigator, though in general the use of zidovudine+lamivudine (300/150mg Combivir®) is recommended. If patients can be included at or before gestational week 20, a 12h pharmacokinetic curve will be recorded at week 20 (± 2 weeks)(Group 1). There should be a minimum of 2 weeks between start of lopinavir and pharmacokinetic recording. If they are included after week 20, the first 12h pharmacokinetic curve will be recorded at gestational week 33 (± 2 weeks)(Group 2). For the patients in both groups a 12 hr curve will be recorded.
  Subjects in Group 1 will be offered to conduct a second 12h pharmacokinetic curve at week 20 (± 2 weeks), but this is only optional. Both groups will be asked to participate in the post partum curve, again this is optional.

SUMMARY:
To determine the pharmacokinetic profile of generic lopinavir/ritonavir tablets To investigate the possible influence of pregnancy and duration of pregnancy To determine the antiviral activity and safety of generic lopinavir/ritonavir® Compare pharmacokinetics parameters before and after pregnancy.

DETAILED DESCRIPTION:
HAART in pregnant HIV-infected serves two goals, preventing mother to child transmission and providing adequate treatment for the mother. Levels of HIV RNA at delivery and the use of antiretrovirals (ARV) are independently associated with decreased transmission[1]. With a HAART regimen the transmission rate can be reduced till under the 2 %[1, 2]. Possibly suitable drugs which can be used during pregnancy is lopinavir/ritonavir based regimens. In Thailand, aluvir is not available therefore a generic lopinavir/ritonavir tablet formulation will be used in our study.

In order to prove adequate levels of lopinavir/ritonavir, we will record 12-hour PK at third trimester. Second trimester and post-partum 12-hour PK are optional. Furthermore, we will collect safety and efficacy throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented positive test for HIV-1 infection
* Subject is at least 18 and not older than 40 years of age at the day of the first dosing of study medication
* Subject is able and willing to sign the Informed Consent Form prior to screening evaluations.
* Pregnant for a maximum of 30 weeks at the day of first dosing of study medication

Exclusion Criteria:

* History of sensitivity/idiosyncrasy to the drug or chemically related compounds or excipients, which may be employed in the trial.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Inability to understand the nature and extent of the trial and the procedures required.
* Abnormal serum transaminases or creatinine, determined as levels being > 3 times upper limit of normal.
* Concomitant use of medications that interfere with Generic lopinavir/ritonavir pharmacokinetics
* Active hepatobiliary or hepatic disease (N.B. chronic hepatitis B/C co-infection is allowed)
* Documented previous virological failure of a lopinavir/ritonavir containing regimen or documented resistance to lopinavir/ritonavir prior to dosing

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetic profile of generic lopinavir/ritonavir tablets 200/50 mg in pregnant Thai HIV-infected women | 1 year

SECONDARY OUTCOMES:
To determine the antiviral activity of generic lopinavir/ritonavir 400/100 mg BID in Thai pregnant women To determine the safety of generic lopinavir/ritonavir® 400/100 mg BID in Thai pregnant women Compare pharmacokinetics parameters before and after | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Surasith Chaithongwongwatthana, MD, Principal Investigator — Department of Obstetrics and Bynecology, Faculty of Medicine, Chulalongkorn University
Locations (1):
- Department of Obsterics and Gynecology, Faculty of Medicine, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- See also: HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org